CLINICAL TRIAL: NCT01495208
Title: This is an Open Label Study to Evaluate the Efficacy of Intravitreal Aflibercept Injection 2mg in Patients With a Persistent FVPED Despite at Least 6 Consecutive Injections With Ranibizumab 0.5 mg
Brief Title: Open Label to Study to Evaluate Effect of Alfilbercept on Patients With (FVPED) Fibrovascular Pigment Epithelial Detachment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVER STUDY
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-05

CONDITIONS: Fibrovascular Pigment Epithelial Detachment
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept (Experimental)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — intravitreal aflibercept injection 2mg

SUMMARY:
This is an open label study to evaluate the efficacy of intravitreal aflibercept injection 2mg in patients with a persistent FVPED despite at least 6 consecutive injections with ranibizumab 0.5 mg.

DETAILED DESCRIPTION:
This is an open label study to evaluate the efficacy of intravitreal aflibercept injection 2mg in patients with a persistent FVPED despite at least 6 consecutive injections with ranibizumab 0.5 mg.

Patients being evaluated at VRM New York with neovascular AMD who have persistent sub-foveal FVPED on OCT despite at least 6 consecutive ranibizumab injections will be considered for the study.

We aim to recruit 25 patients in the study. There have been no statistical tests to calculate sample size; sample size of 25 patients is chosen, making sure that it is feasible financially to conduct the study and logistically to complete the study within 24 weeks. This is a pilot study to assess the effects of intravitreal aflibercept injection on chronic, persistent FVPEDs; currently there is no data regarding visual and anatomical outcomes for this group of patients.

Patients will be reviewed at baseline and then at 4 week intervals (28 ± 7 days). They will receive intravitreal intravitreal aflibercept injection 2mg at each visit. The primary end point of the study is 24 weeks from baseline. Patients who complete the study will have received 6 injections of intravitreal aflibercept injection 2mg.

ELIGIBILITY:
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Subfoveal FVPED assessed using clinical examination and OCT
* Best corrected visual acuity in the study eye between 20 and 85 letters on the ETDRS chart (20/30 to 20/800 Snellen equivalent)
* Prior treatment with at least 6 consecutive injections with ranibizumab 0.5 mg prior to the baseline visit; the last treatment with ranibizumab should not exceed 45 days from the baseline visit.

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation
* Participation in another simultaneous medical investigation or trial
* Prior treatment with ranibizumab therapy in the study eye within 30 days of baseline
* Prior treatment with PDT in the study eye
* Prior intravitreal injection of a corticosteroid (triamcinolone, dexamethasone) within 120 days from baseline.
* Presence of significant subfoveal fibrosis or atrophy determined using SDOCT, fluorescein angiography and clinical examination.
* Presence of fibrous or fibrocellular material occupying more than 50% of the sub-RPE space; assessed using EDI OCT
* Presence of a RPE tear, determined by clinical examination, FA, FAF and OCT
* Intraocular surgery (including cataract surgery) in the study eye within 90 days preceding baseline
* History of pars plana vitrectomy, submacular surgery or any other surgical intervention for vitreo-retinal diseases in the study eye
* Presence of or previous history of diabetic macular edema or proliferative diabetic retinopathy.
* History of uveitis in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment, macular hole and lamellar hole and in the study eye
* Ocular or periocular infection
* Active severe intraocular inflammation
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* In patients with glaucoma, advanced field loss; mean deviation on threshold visual field of more than 12 decibels.
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment.
* History of allergy to fluorescein, ICG or iodine, not amenable to treatment
* Known hypersensitivity to aflibercept or to any of the excipients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in retinal anatomy (size of FVPED, sub-retinal fluid and retinal volume) from baseline; measured using Spectralis OCT (Heidelberg Engineering, Germany) | 24 weeks is the primary end point of the study
  Using the Heidelberg software, subfoveal subretinal fluid (distance between the IS/OS line and the RPE line on SDOCT)
Change in retinal anatomy (size of FVPED, sub-retinal fluid and retinal volume) from baseline; measured using Spectralis OCT (Heidelberg Engineering, Germany) | 24 weeks is the primary end point of the study
  Measure of retinal volume (distance between the ILM and RPE outer margin on SDOCT)
Change in retinal anatomy (size of FVPED, sub-retinal fluid and retinal volume) from baseline; measured using Spectralis OCT (Heidelberg Engineering, Germany) | 24 weeks is the primary end point of the study
  Measure of PED height (distance between ILM and Bruchs membrane (if visible) or the horizontal line where the RPE should be present if it was not elevated)
Change in retinal anatomy (size of FVPED, sub-retinal fluid and retinal volume) from baseline; measured using Spectralis OCT (Heidelberg Engineering, Germany) | 24 weeks is the primary end point of the study
  Measure of maximal diameter of the PED (measured as the point from where the RPE detachment begins to where it ends) will be measured.

SECONDARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) from baseline; measured by ETDRS visual refraction at 4 meters. | 24 weeks is the primary end point of the study
  * Proportion of patients losing ≤ 15 ETDRS letters compared to baseline.
  * Proportion of patients gaining ≥ 5 ETDRS letters compared to baseline.
Mean change in best corrected visual acuity (BCVA) from baseline; measured by ETDRS | 24 weeks is the primary end point of the study
  Measure the Change in sub-RPE tissue characteristics from baseline; determined using EDI-OCT on the Spectralis OCT

CONTACTS AND LOCATIONS:
Overall Officials: Richard Spaide, MD, Principal Investigator — Vitreous -Retina- Macula Consultants of New York
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States